CLINICAL TRIAL: NCT07357584
Title: Efficacy and Safety of Doravirine in the Rapid Initiation of Highly Active Antiretroviral Therapy (HAART) in HIV-1positive Patients Without Prior Treatment
Brief Title: Efficacy and Safety of Doravirine in the Rapid Initiation
Acronym: RapiDO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry); Fundacion IDEAA (Other)
Responsible Party: Principal Investigator, Pedro Enrique Cahn, MD, Fundación Huésped
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-96
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-infection
Keywords: Efficacy; Safety; Doravirine; Rapid initiation of highly active antiretroviral therapy
MeSH Terms: interventions — doravirine; Lamivudine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-randomized, single-arm, non-comparative, open-label study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doravirine /Lamivudine/ Tenofovir Disoproxil (Experimental): Doravirine 100 mg/Lamivudine 300 mg/Tenofovir disoproxilo245 mg
  Interventions: Drug: Doravirine / lamivudine/ Tenofovir Disoproxil Oral Tablet

INTERVENTIONS:
Drug: Doravirine / lamivudine/ Tenofovir Disoproxil Oral Tablet — Pharmaceutical form: Oral tablets Unit dose concentration/dose level(s): 100/300/245 mg Administration instructions: Take one tablet once a day
  Other Names: Delstrigo

SUMMARY:
Protocol title: "Efficacy and safety of doravirine in the rapid initiation of highly active antiretroviral therapy (HAART) in HIV-1positive patients without prior treatment."

DETAILED DESCRIPTION:
Protocol number: FH-96

Primary objective: To evaluate the antiviral activity of DOR/3TC/TDF at week 48 in HIV.

Secondary objectives:

1. To evaluate the antiviral activity of DOR/3TC/TDF at < 200 coIPes/mL at week 48, using the intention-to-treat analysis (FDA snapshot analysis) for the exposed population (ITT-E). 2. To evaluate the antiviral activity of DOR/3TC/TDF at week 48 using an observed analysis (only including patients with available virological data).

3. To evaluate the antiviral activity of DOR/3TC/TDF in the subgroup of participants with baseline ITINN mutations that do not confer resistance to doravirine, (according to the list of mutations defined in the exclusion criteria) by calculating the proportion of patients with viral load <200 coIPes/mL and <50 coIPes/mL at week 48.

4. To evaluate the antiviral activity of DOR/3TC/TDF at <200 coIPes/mL and <50 coIPes/mL at week 24.

5. To evaluate the safety and tolerability of DOR/3TC/TDF. 6. To evaluate the antiviral activity of DOR/3TC/TDF at week 48 in patients with a baseline viral load >100,000 coIPes/mL.

7. Immune response: to evaluate immune recovery (CD4, CD8 and CD4/CD8 T-cell counts at weeks 24 and 48.

8. To evaluate the development of HIV-1 resistance in patients experiencing virological failure while undergoing treatment with DOR/3TC/TDF.

9. To assess changes in weight, BMI, and liIPd profile (total cholesterol, HDL, LDL and triglycerides) at weeks 24 and 48.

Study population: Subjects will be HIV-1 infection patient without ARV experience (naïve) within 30 days of diagnosis, willing to start ARV therapy in a rapid initiation setting, with ≥ 18 years of age, and who meet all inclusion criteria and do not meet any of the exclusion criteria.

Study design: Phase IV, multicenter, non-randomized, single-arm, open-label study describing the antiviral efficacy, safety, and tolerability of DOR/3TC/TDF therapy as rapid initiation therapy in subjects with HIV-1 infection who have not received prior treatment.

Regimens: Doravirine 100 mg; Lamivudine 300 mg; Tenofovir disoproxil 245 mg. Thirteen bottles. (Trade name: DELSTRIGO - MSD). Duration: 48 weeks.

Sample size: 100 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject has to voluntarily signed and dated an informed consent form, approved by an institutional ethics committee.
2. ≥18 years of age.
3. Not previously exposed to ARV (naïve). Subject may have received oral PrEP and PEP within the last 6 months and injectable PrEP and PEP within the last year.
4. Have a received an HIV diagnosis within 30 days prior to selection. Defined as: Having confirmed HIV-1 infection. HIV-1 positive result is considered if the HIV1 RNA in plasma is ≥ 1000 copies/mL or two HIV antibody tests (using two different tests) are positive.

   NOTE: Participants may be included without knowing their baseline viral load. If baseline viral load results are less than 1000 copies/mL, the volunteer's participation will be suspended and they will be considered to have failed the screening test. A viral load brought by the subject may be considered if it was performed within the last 30 days prior to the SCR visit.
5. CD4+ T-cell count: No limit.
6. Subjects able to meet the protocol requirements.

Exclusion Criteria:

1. History of hypersensitivity to doravirine, tenofovir, or lamivudine.
2. Severe hepatic impairment (Child-Pugh C).
3. Active HCV infection requiring specific treatment during study participation at the time of eligibility assessment. If HCV is diagnosed during the study and the participant requires treatment, the decision on whether to continue in the study will be at the investigator's discretion.
4. A woman may be eligible to enter and participate in the study if she is not pregnant (confirmed by a negative urine pregnancy test at the time of screening/baseline). If the baseline visit is scheduled on a different day than the SCR, the urine pregnancy test will be repeated) or breastfeeding and if at least one of the following conditions applies:

   1. Women without reproductive capacity, defined as premenopausal women with tubal ligation or hysterectomy, or documented bilateral oophorectomy; or as postmenopausal women with 12 months of spontaneous amenorrhea, and women ≥ 45 years of age without hormone replacement therapy.
   2. Women with reproductive capacity who agree to adopt one of the contraceptive options in Appendix 2 for at least 30 days after the last dose of study medication and/or completion of the follow-up visit.

   The chosen contraceptive method must be used consistently, according to the approved product label. All study participants must be advised on safer sex practices, including the use of effective barrier methods, and the choice of effective contraceptive method must be documented in the eCRF (Electronic Case Report Form).
5. The subject's general health status, in the investigator's oIPnion, interferes with the requirements of the study.
6. Has a diagnosis of an active opportunistic infection defining AIDS or a malignant neoplasm within 30 days prior to evaluation (except Kaposi's sarcoma with fewer than 10 skin lesions).
7. Is participating or has participated in a clinical study in the last 6 months.
8. Creatinine clearance (CrCl) ≤50 mL/min according to the Cockcroft-Gault equation.
9. Any verified Grade 4 abnormality (except liIPds: HDL, LDL, total cholesterol, triglycerides).
10. History or presence of allergy to study drugs or their components, or to drugs in their class.
11. Subjects taking any medication during the study, including over-the-counter medications and herbal preparations, without the approval of the study physician.
12. Mutations resistant to doravirine, 3TC, or TDF, according to the list described below:

DOR mutations (INNTI):

Doravirine (INNTI) Primary: the presence of one or more ART-resistant mutations will be grounds for exclusion.

Mutations: V106A/M, F227C/V, L234I, Y188L, Y318F, M230I/L. Secondary: the presence of one or more RAMs will be grounds for exclusion. Mutations: A98G, V108I, G190E, H221Y, P225H, F227L, P236L. Others: the presence of five or more RAMs will be grounds for exclusion. Mutations: V90I, L100I, K101E/H/P, K103N/R/S, V106I, I135T, Y181C/I/V, E138A/G/K/Q/R, V170F/T, G190A/Q/S, Y188C/H, F227I, V245E, K311R.

NRTI (TDF) Relevant mutations: Presence of one or more RAM Mutations: K65R, insertion 69, K70R/E, Q151M,

NRTI (3TC) Relevant mutation Presence of IM184V

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-07-13 (Estimated); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Evaluate the antiviral activity of DOR/3TC/TDF at week 48 in HIV patients without prior antiretroviral treatment, in a rapid initiation setting. | 48 Weeks
  Proportion of patients with a viral load < 50 copies/mL at week 48, as determined by an intention-to-treat analysis (FDA snapshot analysis) of the exposed population (ITT-E)

SECONDARY OUTCOMES:
Evaluate the antiviral activity of DOR/3TC/TDF at < 200 copies/mL at week 48, using the intention-to-treat analysis (FDA snapshot analysis) for the exposed population (ITT-E). | 48 Weeks
  Proportion of patients with a viral load < 200 copies/mL at week 48, using intention-to-treat analysis (FDA snapshot analysis) for the exposed population (ITT-E).
Evaluate the antiviral activity of DOR/3TC/TDF at week 48 using an observed analysis (only including patients with available virological data). | 48 Weeks
  Proportion of patients who achieved HIV-1 RNA levels <50 copies/mL at week 48, in those with available data (observed analysis)
Evaluate the antiviral activity of DOR/3TC/TDF in the subgroup of participants with baseline ITINN mutations that do not confer resistance to doravirine, by calculating the proportion of patients with viral load <200 c/mL and <50 c/mL at week 48. | 48 Weeks
  Proportion of patients with viral load < 200 copies/mL and viral load < 50 copies/mL at week 48 in the subgroup of participants with baseline ITINN mutations that do not confer resistance to doravirine, according to the list of mutations defined in the exclusion criteria.
Evaluate the antiviral activity of DOR/3TC/TDF at <200 copies/mL and <50 copies/mL at week 24. | 24 Weeks
  Proportion of patients with viral load < 200 copies/mL and viral load < 50 copies/mL at week 24, using intention-to-treat analysis (FDA snapshot analysis) for the exposed population (ITT-E).
Evaluate the safety and tolerability of DOR/3TC/TDF. | 52 Weeks
  Frequency, type, severity, and seriousness of adverse events and laboratory abnormalities, and proportion of patients who discontinued treatment with DOR/3TC/TDF due to adverse events or death
Evaluate the antiviral activity of DOR/3TC/TDF at week 48 in patients with a baseline viral load >100,000 copies/mL. | 48 Weeks
  Proportion of patients with a baseline HIV-1 RNA level >100,000 c/mL who achieve virological suppression below 50 copies/mL at week 48 (ITT-E analysis).
Immune response: evaluate immune recovery (CD4, CD8 and CD4/CD8 T-cell counts at weeks 24 and 48. | 24 and 48 Weeks
  Changes in CD4 T-cell count, CD8 T-cell count, and CD4/CD8 ratio between baseline and weeks 24 and 48.
Evaluate the development of HIV-1 resistance in patients experiencing virological failure while undergoing treatment with DOR/3TC/TDF | 48 Weeks
  Number and type of resistance mutations in cases of virological failure.
Assess changes in weight and BMI, at weeks 24 and 48. | 24 and 48 Weeks
  Changes in weight and BMI between baseline and weeks 24 and 48. Weight and height will be combined to calculate BMI in kg/m^2. Weight will be measured at all visits and height only at the baseline visit.
Assess changes in lipid profile (total cholesterol, HDL, LDL and triglycerides) at weeks 24 and 48. | 24 and 48 Weeks
  Changes in lipid profile (total cholesterol, HDL, LDL and triglycerides) between baseline and weeks 24 and 48.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Fundacion IDEAA -Infectologia de atencion ambulatoria, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Fundacion Huesped, Buenos Aires

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared upon request, 6 months after last patient´s last visit. URL not yet available.